CLINICAL TRIAL: NCT00836485
Title: A Prospective, Multi-Center, Double-Masked, Randomized, Placebo-Controlled Evaluation of the Safety and Efficacy of Ketotifen 4.0% Patch as Compared to Placebo Patch, Olopatadine 0.2% Ophthalmic Solution, and Artificial Tears in the Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis
Brief Title: Evaluation of the Safety and Efficacy of Ketotifen 4.0% Patch as Compared to Placebo Patch, Olopatadine 0.2% Ophthalmic Solution, and Artificial Tears in the Conjunctival Allergen Challenge (CAC) Model of Acute Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Senju USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNJ-ALK201/08-003-11
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen; Transdermal Patch; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Ketotifen 4.0% Patch
  Interventions: Drug: Ketotifen 4.0% Patch
- 2 (Placebo Comparator): Placebo Patch
  Interventions: Drug: Placebo
- 3 (Active Comparator): Pataday(TM)
  Interventions: Drug: Olopatadine 0.2%
- 4 (Placebo Comparator): Placebo eye drops
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Ketotifen 4.0% Patch — This investigational drug is a transdermal patch indicated to treat allergic conjunctivitis. Application is intended for overnight wear between 8-10 hours.
  Arms: 1
Drug: Placebo — The control is a placebo patch that contains only the inactive ingredients of ketotifen.
  Arms: 2
Drug: Olopatadine 0.2% — 1 gtt/eye on two separate occasions
  Other Names: Pataday(TM)
  Arms: 3
Drug: Artificial tears — 1 gtt/eye on two separate occasions
  Arms: 4

SUMMARY:
This is a phase 2 study that will consist of 4 visits over a 5 week period. Drug will be evaluated using the conjunctival allergen challenge model of allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age of either sex and any race
* positive history of ocular allergies and a positive skin test reaction to cat hair, cat dander, dog dander, grasses, ragweed, trees, dust mites, and/or cockroaches within the past 24 months
* able and willing to avoid all disallowed medication for the washout period and during the study

Exclusion Criteria:

* active ocular infection or skin condition
* ocular surgery within the past 3 months
* pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Ocular itching and bulbar conjunctival redness | Visit 3 and Visit 4

SECONDARY OUTCOMES:
Ocular: Ciliary, episcleral, and inferior palpebral conjunctival redness; chemosis; lid swelling; tearing; ocular mucous discharge | Visit 3 and Visit 4
Nasal: Rhinorrhea; ear or palate pruritis; nasal pruritis; nasal congestion; and a composite score of all nasal symptoms | Visit 3 and Visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — ORA, Inc.; TBD TBD, Principal Investigator
Locations (1):
- Ora, Andover, Massachusetts, United States